CLINICAL TRIAL: NCT03130816
Title: Mechanism of Allogeneic Umbilical Cord Blood Therapy in Cerebral Palsy
Brief Title: Mechanism of Allogeneic UCB Therapy in Cerebral Palsy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, MinYoung Kim, MD, PhD, Professor, Bundang CHA Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-06-093
Record Dates: First submitted 2017-04-20; First posted 2017-04-27 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Cerebral Palsy; Child Development
Keywords: Umbilical cord blood transplantation; Cytokine changes
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with cerebral palsy volunteered for participation in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- allogeneic cord blood transplantation (Experimental): Intravenous(IV) infusion will be done by the following method A. After 4 hours of fasting, subjects will be sedated with chloral hydrate (Pocral®) syrup B. Intravenous infusion will be conducted in stem cell center, CHA Bundang Medical Center and the therapy will be performed by the Principal Investigator or a physician delegated from the Principal Investigator. The physician conducting the infusion will not participate in the efficacy and result analysis of this study.
  C. Oxygen saturation will be monitored during therapy.
  Interventions: Biological: allogeneic cord blood transplantation

INTERVENTIONS:
Biological: allogeneic cord blood transplantation — UCB with total nucleated cell count ≤ 7x108/kg will be used for this clinical trial. Suitable UCB (i.e., containing total nucleated cell count ≥2x107/kg with three or less mismatch among HLA-A, -B, and -DR) will be selected. This criterion was selected upon the rationale that even though minimal HLA mismatch is preferred, prior studies indicate significant effects of UCB therapy for patients with 3 HLA mismatches.

SUMMARY:
In our prior study on the therapeutic mechanism of UCB, changes in cytokine levels were observed but the results are inconclusive and further studies on animal models and changes of protein expression before and after UCB therapy in the clinical settings are required.

The changes in protein expression will be assessed by multiplex RT-PCR mRNA assay. Clinical efficacy of UCB therapy will be evaluated with various functional assessment tools. Factors regarding UCB therapy (number of transplanted cells, HLA matching status, serum level of immunosuppressant, etc.) and patient factors (age, functional status, etc.) will be analyzed for correlation with protein expression after UCB therapy. Several target proteins for analysis are available. Pentraxin and toll-like receptor (TLR) 4 are receptors modulating intrinsic immune reaction and was shown to have a significant correlation with clinical efficacy of stem cell therapy. Ubiquitine is a regulatory protein that combines with the target protein and affects its degradation, interaction, localization and activation. The ubiquitine system controls total protein quantity for homeostasis and can be found in all tissues. Deubiquitination (DUB) enzyme down-regulates this ubiquitine and is known to modulate all cellular changes

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with cerebral palsy
2. Age of ≥10 months and ≤20 years
3. Mismatch in HLA-A, B, and DR ≤3, and total nucleated cell count ≥2x107/kg. If the cell count is less than given values, more than 2 units may be used.
4. Voluntary decision to participation in the study with informed consent agreed and obtained from the subject's representative.
5. Patient and/or representatives are both willing and capable of being hospitalized according to the schedule specified in the protocol and continue the study for 12 months after study entry.
6. If the patient has participated in another clinical trial, at least 3 months should have passed since end of the study.

Exclusion Criteria:

1. Current aspiration pneumonia
2. Known genetic disease
3. History of hypersensitivity reaction to any study drugs pertinent to the study
4. Patient with severe convulsion disease who has clinical convulsion despite combination therapy with 3 or more agents
5. Uncontrolled hypertension defined as systolic blood pressure >115 mmHg and/or diastolic blood pressure >70 mmHg
6. Hepatic impairment defined as asparate aminotransferase (AST) >55 IU/L and/or alanine aminotrasferase (ALT) >45 IU/L
7. Renal impairment defined as creatinine (Cr) ≥1.3 mg/dL
8. Presence of diagnosed or suspected malignant tumor and/or hematologic malignancy
9. Non-compliance with study visits specified in the protocol or poor compliance of care-giver.
10. Any factors not specified above that the principal investigator determines medically inadequate for participation in this study.

Ages: 10 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-07-29 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-05-21 (Actual)

PRIMARY OUTCOMES:
Change of GMFM | Baseline before UCB administration, months 3, 6, and 12 after UCB treatment
  Gross motor function measure measured at baseline before UCB administration is compared to the score measured at months 3, 6, and 12 after UCB treatment.

SECONDARY OUTCOMES:
Change of mRNA assay | Change between the baseline level before UCB therapy and levels after UCB administration at 2 days, 1 week, 5 weeks, and 12 months
  Separate peripheral blood mononuclear cell (PBMC) from the patients' blood sample and screen for changes in protein enzymes including those related to DUB at the mRNA level after UCB therapy.
Change of GMPM | Baseline before UCB administration, months 3, 6, and 12 after UCB treatment
  Dissociated Movement, Coordination, Alignment, Weight shift, and Stability are rated with GMPM (Gross Motor Performance Measure). Each raw score (1-5 point) and converted percent scores are evaluated. Total score is 100(%), higher scores indicate better function. GMPM measured at baseline before UCB administration is compared to the score measured at months 3, 6, and 12 after UCB treatment.

CONTACTS AND LOCATIONS:
Overall Officials: MinYoung Kim, MD, PhD, Principal Investigator — CHA University
Locations (1):
- CHA Bundang Medical Center, Seongnam, Gyeonggido, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Suh MR, Min K, Cho KH, Kim J, Lim I, Park M, Noh EM, Kim MY. Maintenance of the synergistic effects of cord blood cells and erythropoietin combination therapy after additional cord blood infusion in children with cerebral palsy: 1-year open-label extension study of randomized placebo-controlled trial. Stem Cell Res Ther. 2023 Dec 12;14(1):362. doi: 10.1186/s13287-023-03600-4. PMID 38087394